CLINICAL TRIAL: NCT07006532
Title: Treatment of Chronic Active Antibody Mediated Rejection in Kidney Transplant Recipients With Tocilizumab ,IVIG, Plasmapheresis, Rituximab Versus IVIG, Plasmapheresis , Rituximab
Brief Title: Treatment of Chronic Active Antibody Mediated Rejection With Tocilizumab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, assistant professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBMU-1404-2/2
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Plasmapheresis plus Rituximab plus IVIG
- Intervention (Other): Standard of care plus Tocilizumab
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — The trial is an open-labeled randomized clinical trial that evaluates the safety and efficacy of Tocilizumab as an add-on therapy to standard of care treatment of Plasmapheresis, IVIG, and Rituximab in treatment of CAMR in kidney transplant recipients.
  Arms: Intervention

SUMMARY:
Chronic active antibody mediated rejection (CAMR) is a therapeutic challenge in transplant recipients that does not respond well to conventional treatments for acute antibody mediated rejection (AMR). Annually, 5000 kidney transplants are lost in the United States due to CAMR. The two-year graft survival rate in CAMR is approximately 20%, highlighting the need for a more efficient therapy for CAMR and directly targeting donor specific antibody (DSA) producing cells and reducing CAMRThere is no established treatment for this problem. While many centers intensify and optimize the dosage of immunosuppressive drugs, treatments such as plasmapheresis, IVIG, and rituximab, although effective in treating AMR, have not been successful in reducing DSA or improving kidney graft survival in CAMR patients. Despite these treatments, two-year graft survival can increase up to 55%. The use of anti-plasma cell treatments like bortezomib has also yielded inconsistent results.

DETAILED DESCRIPTION:
The trial is an open-labeled randomized clinical trial that evaluates the safety and efficacy of Tocilizumab as an add-on therapy to standard of care treatment of Plasmapheresis, IVIG, and Rituximab in treatment of CAMR in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. eGFR> 25 cc/min
3. Chronicity index <8
4. IFTA<40%
5. EBV IgG positive

Exclusion Criteria:

1. Active or recurrent infections
2. History of malignancy, unless in remission for more than 2 years with no relapse
3. abnormal liver function tests
4. Platelet < 100,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
GFR | through study completion, an average of 1 year
  cc/min/1.73 m

CONTACTS AND LOCATIONS:
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No